CLINICAL TRIAL: NCT05535049
Title: The Effect of Non-surgical Periodontal Treatment on Serum and Gingival Crevicular Fluid Periostin Levels
Brief Title: Non-surgical Periodontal Treatment and Periostin Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Aysegul SARI, Scientific research projects, Mustafa Kemal University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019/118
Record Dates: First submitted 2022-09-06; First posted 2022-09-10 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Periodontal Treatment, Cytokines
Keywords: Periodontitis; Periostin; Periodontal treatment; Gingival crevicular fluid
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periodontally healthy group (No Intervention): 24 participants were included in this group.
- Periodontitis group (Active Comparator): 24 participants were included in this group.
  Interventions: Procedure: Non-surgical periodontal treatment

INTERVENTIONS:
Procedure: Non-surgical periodontal treatment — Full month non-surgical periodontal treatment procedure was applied to the periodontitis group.
  Arms: Periodontitis group

SUMMARY:
Two different studies were planned from the recruited samples. The aim of these studies was to investigate the effect of non-surgical periodontal treatment on the inflammatory markers levels in serum and gingival crevicular fluid (GCF) in patients with periodontitis.

There were two groups consisting of individuals who had periodontitis and those who were healthy, with 24 individuals in each group.

Periostin levels were assessed at baseline, at the 24th h, 48th h, 14th day 1st month, 3rd month after non-surgical periodontal treatment in serum and GCF samples by the Elisa method in the first study. In parallel, interleukin 1 (IL)-beta and fibroblast growth factor levels were measured.

Progranulin levels were assessed at baseline, at the 24th h, 48th h, 14th day 1st month, 3rd month after non-surgical periodontal treatment in serum and GCF samples by the Luminex method in the second study. In parallel, vascular endothelial growth factor, IL-1 beta, tumor necrosis factor-alpha, and IL-10 levels were measured.

DETAILED DESCRIPTION:
The First Study

The observational prospective study was designed to characterize periostin changes over time after non-surgical periodontal treatment in serum and GCF in the Department of Periodontology in the Faculty of Dentistry at Hatay Mustafa Kemal University, Hatay, Turkey. The study protocol was approved by the Ethics Committee for the Use of Human Subjects in Research of Hatay Mustafa Kemal University (Protocol No: 2019/118). The study was carried out in accordance with the tenets of the Declaration of Helsinki and conducted in CONSORT guidelines (Schulz, Altman, & Moher, 2010). This study project was financially supported by Hatay Mustafa Kemal University Scientific Research Projects Coordinator (19M051).

Individuals were included in the study from December 2019 through August 2021. Written informed consent was obtained from each participant before the clinical periodontal examination.

Study Population

Forty-eight adult individuals were enrolled in the study. Participants were recruited into 2 sex matched groups with 24 participants in each: periodontally healthy (PH) and periodontitis (P) groups. In accordance with the demographic variables of the patients included in the P group, the patients in the PH groups were included.

Periodontal Parameters

Periodontal clinical parameters were recorded by a single calibrated examiner (k =0.95) (author AS). Intra-examiner agreement was determined for CAL. The intra-examiner reproducibility was determined through repeated examinations of 10 subjects with a one-hour interval. Clinical periodontal measurements were assessed using the following periodontal measurements for periodontal diagnosis in both groups and also at the 1st month, 3rd month after non-surgical periodontal treatment in the periodontitis group.

The measurements were performed using a Williams periodontal probe (Hu-Friedy, Chicago, IL, USA) and included probing pocket depth (PPD), clinical attachment level (CAL), plaque index (PI) (Silness & Loe, 1964), gingival index (GI) (Loe & Silness, 1963), and percentage bleeding on probing (BOP) (Ainamo & Bay, 1975) at six sites per tooth (mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual and disto-lingual) on each tooth.

Diagnosis of periodontal diseases and conditions was made according to the radiographic and clinical diagnostic criteria proposed by the 2017 World Workshop on Classification of Periodontal and Peri-implant Diseases and Conditions (Caton et al., 2018). Individuals with BOP < 10% without attachment loss and radiographic bone loss were considered to have periodontal health (Tonetti & Sanz, 2019). The criteria for periodontitis included patients with CAL ≥ 5 mm in two or more interproximal sites and PPD ≥ 6 mm in one or more interproximal sites. Only stage III-IV (severe) periodontitis was included in the present study (Tonetti, Greenwell, & Kornman, 2018).

Periodontal Intervention

Periodontitis patients were treated by one-stage full-mouth disinfection. Full-mouth disinfection included full-mouth scaling and root planning procedures within 24 h in two sessions. Each session was practiced for 60 min on two consecutive days. Subgingival irrigation and tongue brushing were made with 1% CHX gel for 1 min. Mouthwashes with 0.12% CHX were performed for 30 s at the beginning and at the end of each session and twice a day for 2 weeks (Quirynen et al., 1995).

Collection of GCF Samples

GCF samples were collected following 8 hours of night fasting and one week after clinical periodontal measurements at baseline in two groups and then at the the 24th h, 48th h, 14th day 1st month, 3rd month after non-surgical periodontal treatment (Akalin, Baltacioglu, Alver, & Karabulut, 2007). The samples were collected from the teeth side with PPDs ≥6 mm, and BOP positive in patients with periodontitis. Six GCF samples were taken per participant. Samples were collected from a mesial and a distal site on each of three teeth (incisors, premolars, and molars). Saliva contamination was prevented by isolation with cotton rolls and gently air-drying the sampling area. Samples contaminated with saliva or blood were not included. Plaque was gently removed from the sampling area by the periodontal curette. The samples were collected within 30 seconds with standardized paper strips (Periopaper; Oraflow Inc., Plainview, NY) by the orifice method.(Rudin, Overdiek, & Rateitschak, 1970) The volumes were measured on a pre-calibrated electronic gingival fluid measuring device (Oraflow Inc., Plainview, NY)|| (Chapple, Landini, Griffiths, Patel, & Ward, 1999). The values of the electronic device were referenced to a standard curve and converted to an actual volume (µl). All of the Periopaper strips were pooled in plastic Eppendorf microcentrifuge tubes. They were stored at -80 °C until the biochemical analysis.

All samples were thawed and 375 μl of phosphate buffered saline (pH:7.00, 10 mM Na2PO4, 137 mM NaCl, and 2.7 mM KCl) was added into the eppendorf tubes containing the sample strips. Subsequently, samples were eluted for 30 minutes at room temperature and (Chapple et al., 1997) centrifuged at 11000×g for 15 min at 4 °C. The measurement of periostin, IL-1β, and FGF levels were assayed.

Collection of Serum Samples

Peripheral venous blood samples were taken from the patients. The serum was separated from the cells by centrifugation at 2000 rpm for 10 min, after which it was stored at -80°C, until the biochemical analysis was performed.

Laboratory Analyses

Periostin, IL-1β, and FGF levels were measured by the enzyme-linked immunosorbent assay (ELISA) using commercially available kits at 450 nm wavelength in ELISA Reader (Thermo Fisher Scientific Multiscan Go-Finland).

Measurement of periostin levels in GCF samples

Periostin levels were measured by ELABSCIENCE Human POSTN/OSF-2 (Kit Cat No: E-EL-H6113). The assay ranges for the periostin were 3.13-200 ng/ml; sensitivity, 1.88 ng/ml, intra and inter assay coefficients of variance (CV%) were < 10%.

Measurement of IL-1β levels in GCF samples

IL-1β levels were measured by ELABSCIENCE Human IL-1β (Kit Cat No: E-EL-H0149). The assay ranges for the IL-1β were 7.81-500 pg/ml; sensitivity, 4.69 pg/ml, intra and inter assay coefficients of variance (CV%) were < 10%.

Measurement of FGF levels in GCF samples

FGF levels were measured by ELABSCIENCE Human FGF21 (Kit Cat No: E-EL-H0074). The assay ranges for the FGF were 31.25-2000 pg/ml; sensitivity, 18.75 pg/ml, intra and inter assay coefficients of variance (CV%) were < 10%.

The Second Study

The study aimed to evaluate the effect of non-surgical periodontal treatment on serum and gingival crevicular fluid progranulin levels.

3 paper strips and serum samples for each patient recruited from the same patients and same methods as back-up samples were transferred to King's College London Dental Institute, Periodontology Unit, Centre for Host-Microbiome Interactions, London, UK; after a material transfer agreement signed between Hatay Mustafa Kemal University, Hatay, Turkey and King's College London, London, UK in May 2022 for another study. T The study protocol was approved by the Ethics Committee for the Use of Human Subjects in Research of Hatay Mustafa Kemal University (Protocol No: 2022/90). The study was carried out in accordance with the tenets of the Declaration of Helsinki and conducted in the CONSORT guidelines (Schulz, Altman, & Moher, 2010). This study project was financially supported by King's College London internal departmental funds.

GCF Samples Elution

50 μL of PBS/protease inhibitor cocktail (PBS with protease inhibitors 1X, Complete ULTRA tablets, Mini; EDTA-free) were added to a sterile microcentrifuge tube included 3 paper strips and centrifuged at 11000 rpm for 15 min at 4 C for GCF elutiation. This procedure was repeated two times and obtained a total volume of 100 μL. They were stored at -80 °C until the biochemical analysis.

Serum and GCF Samples Analyses

Luminex bead-based multiplex immunoassay (Luminex, R&D systems, Minneapolis, MN) was used to carry out the analysis (in duplicate) of each sample. A custom-made 5-plex kit included inflammatory and regenerative markers: Progranulin (PGRN), VEGF, interleukin (IL)-1 beta, tumor necrosis factor-alpha (TNF-alfa), and IL-10.

Each 50-μL sample was resuspended in a dedicated well with a microparticle cocktail of antibodies covered with a foil plate sealer on magnetic beads and incubated for 2 h on a horizontal orbital microplate shaker. Following washes, the biotin antibody cocktail was added and incubated for 1 h as previously reported. After the washes, streptavidin-phycoerythrin (Streptavidin-PE) incubation was carried out for 30 min. Then, the samples were put into the Luminex MAGPIX analyzer (Luminex; R&D systems) to read. The marker values were obtained as pg/mL.

Statistical Analysis

The normality of the distribution of continuous variables was tested by the Shapiro-Wilk test. Descriptive statistics were presented as mean and standard deviation (mean±sd) for parametric distributed variables and median (interquartile range) for the non-parametric distributed variables.

The chi-square test was used to analyze the associations between categorical variables. The Student t-test for normally distributed numerical variables and Mann Whitney u test for non-normally distributed numerical variables were performed to compare 2 independent groups for numerical data. Freidman test was performed for different time points with non-parametric variables. Dunn multiple comparison tests were performed for post hoc pairwise multiple comparison analyses.

Statistical analysis was performed with SPSS for Windows version 24.0 and P value <0.05 was accepted as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* individuals who had never smoked;
* individuals who had no history of periodontal treatment in the past 6 months;
* individuals who had had no antibiotic therapy in the past 3 months;
* individuals who had more than 18 teeth.

Exclusion Criteria:

* individuals who were pregnant;
* individuals were current or former smokers;
* individuals who had any self-reported systemic condition or disease, which are confounding factors e.g. AIDS, rheumatoid arthritis, cardiovascular diseases, diabetes.

Ages: 24 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of Periostin levels in non-surgical periodontal treatment | 0-3 month
  The effect of non-surgical periodontal treatment on serum and gingival crevicular fluid periostin levels

SECONDARY OUTCOMES:
Evaluation of IL-1B and FGF levels in non-surgical periodontal treatment | 0-3 month
  The effect of non-surgical periodontal treatment on serum and gingival crevicular fluid cytokines levels

CONTACTS AND LOCATIONS:
Overall Officials: Aysegul Sari, PhD, Principal Investigator — Hatay Mustafa Kemal University Dental Faculty; Oguzhan Ozcan, Prof, Study Chair — Hatay Mustafa Kemal University Medical Faculty; Alpdogan Kantarci, Prof, Study Director — Boston University Goldman School of Dental Medicine
Locations (1):
- Mustafa Kemal University, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ainamo J, Bay I. Problems and proposals for recording gingivitis and plaque. Int Dent J. 1975 Dec;25(4):229-35. PMID 1058834
- [Result] Caton JG, Armitage G, Berglundh T, Chapple ILC, Jepsen S, Kornman KS, Mealey BL, Papapanou PN, Sanz M, Tonetti MS. A new classification scheme for periodontal and peri-implant diseases and conditions - Introduction and key changes from the 1999 classification. J Periodontol. 2018 Jun;89 Suppl 1:S1-S8. doi: 10.1002/JPER.18-0157. PMID 29926946
- [Result] Chapple IL, Landini G, Griffiths GS, Patel NC, Ward RS. Calibration of the Periotron 8000 and 6000 by polynomial regression. J Periodontal Res. 1999 Feb;34(2):79-86. doi: 10.1111/j.1600-0765.1999.tb02226.x. PMID 10207836
- [Result] Chapple IL, Mason GI, Garner I, Matthews JB, Thorpe GH, Maxwell SR, Whitehead TP. Enhanced chemiluminescent assay for measuring the total antioxidant capacity of serum, saliva and crevicular fluid. Ann Clin Biochem. 1997 Jul;34 ( Pt 4):412-21. doi: 10.1177/000456329703400413. PMID 9247675
- [Result] LOE H, SILNESS J. PERIODONTAL DISEASE IN PREGNANCY. I. PREVALENCE AND SEVERITY. Acta Odontol Scand. 1963 Dec;21:533-51. doi: 10.3109/00016356309011240. No abstract available. PMID 14121956
- [Result] Quirynen M, Bollen CM, Vandekerckhove BN, Dekeyser C, Papaioannou W, Eyssen H. Full- vs. partial-mouth disinfection in the treatment of periodontal infections: short-term clinical and microbiological observations. J Dent Res. 1995 Aug;74(8):1459-67. doi: 10.1177/00220345950740080501. PMID 7560400
- [Result] Rudin HJ, Overdiek HF, Rateitschak KH. Correlation between sulcus fluid rate and clinical and histological inflammation of the marginal gingiva. Helv Odontol Acta. 1970 Apr;14(1):21-6. No abstract available. PMID 5438796
- [Result] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomized trials. Ann Intern Med. 2010 Jun 1;152(11):726-32. doi: 10.7326/0003-4819-152-11-201006010-00232. Epub 2010 Mar 24. PMID 20335313
- [Result] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464
- [Result] Tonetti MS, Greenwell H, Kornman KS. Staging and grading of periodontitis: Framework and proposal of a new classification and case definition. J Clin Periodontol. 2018 Jun;45 Suppl 20:S149-S161. doi: 10.1111/jcpe.12945. PMID 29926495
- [Result] Tonetti MS, Sanz M. Implementation of the new classification of periodontal diseases: Decision-making algorithms for clinical practice and education. J Clin Periodontol. 2019 Apr;46(4):398-405. doi: 10.1111/jcpe.13104. PMID 30883878
- [Result] Yang N, Li Y, Wang G, Ding Y, Jin Y, Xu Y. Tumor necrosis factor-alpha suppresses adipogenic and osteogenic differentiation of human periodontal ligament stem cell by inhibiting miR-21/Spry1 functional axis. Differentiation. 2017 Sep-Oct;97:33-43. doi: 10.1016/j.diff.2017.08.004. Epub 2017 Sep 1. PMID 28946056
- [Result] Daniel R, He Z, Carmichael KP, Halper J, Bateman A. Cellular localization of gene expression for progranulin. J Histochem Cytochem. 2000 Jul;48(7):999-1009. doi: 10.1177/002215540004800713. PMID 10858277
- [Result] Li X, Zuo Z, Chen Q, Li J, Tang W, Yang P. Progranulin is highly expressed in patients with chronic periodontitis and protects against experimental periodontitis in rats. J Periodontol. 2018 Dec;89(12):1418-1427. doi: 10.1002/JPER.18-0132. Epub 2018 Sep 11. PMID 29999528
- [Result] Horiuchi K, Amizuka N, Takeshita S, Takamatsu H, Katsuura M, Ozawa H, Toyama Y, Bonewald LF, Kudo A. Identification and characterization of a novel protein, periostin, with restricted expression to periosteum and periodontal ligament and increased expression by transforming growth factor beta. J Bone Miner Res. 1999 Jul;14(7):1239-49. doi: 10.1359/jbmr.1999.14.7.1239. PMID 10404027
- [Result] Matsuzawa M, Arai C, Nomura Y, Murata T, Yamakoshi Y, Oida S, Hanada N, Nakamura Y. Periostin of human periodontal ligament fibroblasts promotes migration of human mesenchymal stem cell through the alphavbeta3 integrin/FAK/PI3K/Akt pathway. J Periodontal Res. 2015 Dec;50(6):855-63. doi: 10.1111/jre.12277. Epub 2015 Apr 20. PMID 25900259
- [Derived] Sari A, Santamaria P, Nibali L. The effect of non-surgical periodontal treatment on progranulin levels. J Periodontol. 2025 Aug 25. doi: 10.1002/jper.11396. Online ahead of print. PMID 40853679